CLINICAL TRIAL: NCT02255695
Title: Effects of a School-based Exercise Program on Posture, Trunk Range of Motion, and Musculoskeletal Pain - A Randomized, Controlled Trial
Brief Title: Effects of a School-based Exercise Program on Posture, Trunk Range of Motion, and Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Mariana Vieira Batistão, Master, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 472552/2010-4
Record Dates: First submitted 2014-07-24; First posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Musculoskeletal and Connective Tissue Disorders
Keywords: posture; child; prevention; muscle strength; muscle stretching exercises; exercise therapy; disease management; musculoskeletal pain; adolescent; spinal curvatures
MeSH Terms: conditions — Connective Tissue Diseases; Musculoskeletal Pain; Spinal Curvatures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Control group
- School-based exercise program (Experimental): School-based exercise program
  Interventions: Other: School-based exercise program

INTERVENTIONS:
Other: School-based exercise program — The exercise program was applied, twice a week, for 8 weeks, with sessions of 50 minutes, in groups of 10 students. The exercise program was elaborate to restore muscular balance through flexibility, endurance and muscular strength. To promote flexibility stretching exercises for rotator neck muscles, lateral neck flexors, levator scapulae, upper trapezius, erector spinae, major and minor pectoralis, rhomboids, spinal lateral flexors, column rotators, piriformis, hamstrings, quadriceps, hip adductors and abductors were applied. Strengthening exercises were applied for the development of strength, endurance and control of deep flexor muscles of the cervical spine, stabilizers of the glenohumeral joint and scapula, abdominals, spine extensors and hip extensors.
  Other Names: Exercise group; Intervention group; Program based on stretching and strengthening exercises
  Arms: School-based exercise program

SUMMARY:
The objective of this study was to evaluate the effects of a school-based exercise program on posture, trunk range of motion and musculoskeletal pain in schoolchildren. This study was a Randomized controlled trial. The hypothesis was that the exercise group would have the postural deviations corrected, would have the trunk range of motion increased and would have the prevalence of pain decreased, while the control group would have not. Three schools from Brazil participated. The students that have been included (n=300) were randomly allocated to experimental (EG) or control group (CG). The intervention for EG consisted in a program based on stretching and strengthening exercises, applied twice a week, for eight weeks, with group sessions of 50 minutes. CG did not perform any intervention. Qualitative and quantitative postural evaluation (PAS/SAPO), musculoskeletal pain (self-report) and trunk mobility were collected.

ELIGIBILITY:
Inclusion Criteria: to attend elementary school and deliver the consent term signed by the parents.

-

Exclusion Criteria: presence of disability on musculoskeletal or neurological system, exercise intolerance or attendance less than 50% in the exercise sections

-

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2008-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Changes in the qualitative postural assessment from the baseline | Two time points: baseline and 9 weeks
  Qualitative postural assessment was performed by a physiotherapist through the photographic records. The photos were recorded with the students in swimsuits and no shoes. The subject was positioned over the gyratory platform to avoid reposition for the photographic record, besides the plumb line, with the feet lined and separated by hip width. The records were performed in the frontal and sagittal planes, in the anterior, posterior and lateral view. According to the positioning of the structures in relation to the plumb line, the presence of postural changes was classified by the physiotherapist. Lateral tilt and forward head, shoulder protrusion, cervical lordosis, thoracic kyphosis, and lumbar lordosis were evaluated.

SECONDARY OUTCOMES:
Changes in the quantitative postural assessment from the baseline | Two time points: baseline and 9 weeks
  Postural Assessment Software (PAS/SAPo) was used to quantitatively assess posture. Reflective markers were placed by a trained physiotherapist on the anatomical landmarks of the subject. The subject was positioned over the gyratory platform, and photographic records were performed in the frontal and sagittal planes, in the anterior, posterior and lateral view.
  The analysis followed the guidelines of PAS/SAPo. The photos were aligned and calibrated. The reflective markers were identified and the protocol of measures of the PAS/SAPo was used, providing the following parameters: horizontal alignment of the acromions, horizontal alignment of the ASIS, angle between acromions and ASIS, vertical alignment of the trunk, horizontal alignment of the pelvis, horizontal alignment of the head, vertical alignment of the head.
Changes in trunk range of motion from baseline | Two time points: baseline and 9 weeks
  A photogrammetric technique was used to measure the trunk flexion angle. This angle is formed between the line joining the markers attached on anterior superior iliac spine (ASIS) and greater trochanter and the line joining the marker fixed on the spinous process of the C7 vertebra and the one fixed on the ASIS. Two photographs were recorded; one in the upright position and the other in maximum trunk flexion. The trunk mobility was estimated by the difference between the values obtained in the two photographs. This procedure was performed in PAS/SAPo software.
Changes in the prevalence of musculoskeletal pain from baseline | Two time points: baseline and 9 weeks
  The presence of pain was evaluated by self-report. The Nordic Questionnaire of Musculoskeletal Symptoms body map was used to provide pain localization and data from musculoskeletal pain during the last 7 days. The pain intensity was also investigated by asking to the children about their pain in a 11-point scale, in which 0 is lack of pain and 10 is the greatest pain that the children had ever experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana V Batistão, Master, Principal Investigator — Universidade Federal de Sao Carlos; Tatiana O Sato, Doctorade, Study Director — Universidade Federal de Sao Carlos
Locations (1):
- Universidade Federal de São Carlos, São Carlos, São Paulo, Brazil

REFERENCES:
- [Background] Cardon G, Balague F. Low back pain prevention's effects in schoolchildren. What is the evidence? Eur Spine J. 2004 Dec;13(8):663-79. doi: 10.1007/s00586-004-0749-6. Epub 2004 Jun 15. PMID 15662541
- [Background] Hakala P, Rimpela A, Salminen JJ, Virtanen SM, Rimpela M. Back, neck, and shoulder pain in Finnish adolescents: national cross sectional surveys. BMJ. 2002 Oct 5;325(7367):743. doi: 10.1136/bmj.325.7367.743. PMID 12364301
- [Background] Limon S, Valinsky LJ, Ben-Shalom Y. Children at risk: risk factors for low back pain in the elementary school environment. Spine (Phila Pa 1976). 2004 Mar 15;29(6):697-702. doi: 10.1097/01.brs.0000116695.09697.22. PMID 15014281
- [Background] van Gent C, Dols JJ, de Rover CM, Hira Sing RA, de Vet HC. The weight of schoolbags and the occurrence of neck, shoulder, and back pain in young adolescents. Spine (Phila Pa 1976). 2003 May 1;28(9):916-21. doi: 10.1097/01.BRS.0000058721.69053.EC. PMID 12942008
- [Background] Coleman J, Straker L, Ciccarelli M. Why do children think they get discomfort related to daily activities? Work. 2009;32(3):267-74. doi: 10.3233/WOR-2009-0825. PMID 19369719
- [Background] Juskeliene V, Magnus P, Bakketeig LS, Dailidiene N, Jurkuvenas V. Prevalence and risk factors for asymmetric posture in preschool children aged 6-7 years. Int J Epidemiol. 1996 Oct;25(5):1053-9. doi: 10.1093/ije/25.5.1053. PMID 8921494
- [Background] Hrysomallis C, Goodman C. A review of resistance exercise and posture realignment. J Strength Cond Res. 2001 Aug;15(3):385-90. PMID 11710670
- [Background] Kjaer P, Leboeuf-Yde C, Sorensen JS, Bendix T. An epidemiologic study of MRI and low back pain in 13-year-old children. Spine (Phila Pa 1976). 2005 Apr 1;30(7):798-806. doi: 10.1097/01.brs.0000157424.72598.ec. PMID 15803084
- [Background] Correa EC, Berzin F. Efficacy of physical therapy on cervical muscle activity and on body posture in school-age mouth breathing children. Int J Pediatr Otorhinolaryngol. 2007 Oct;71(10):1527-35. doi: 10.1016/j.ijporl.2007.05.031. Epub 2007 Jul 30. PMID 17659787
- [Background] Zaina F, Atanasio S, Ferraro C, Fusco C, Negrini A, Romano M, Negrini S. Review of rehabilitation and orthopedic conservative approach to sagittal plane diseases during growth: hyperkyphosis, junctional kyphosis, and Scheuermann disease. Eur J Phys Rehabil Med. 2009 Dec;45(4):595-603. PMID 20032919
- [Background] Ahlqwist A, Hagman M, Kjellby-Wendt G, Beckung E. Physical therapy treatment of back complaints on children and adolescents. Spine (Phila Pa 1976). 2008 Sep 15;33(20):E721-7. doi: 10.1097/BRS.0b013e318182c347. PMID 18794746
- [Background] Fanucchi GL, Stewart A, Jordaan R, Becker P. Exercise reduces the intensity and prevalence of low back pain in 12-13 year old children: a randomised trial. Aust J Physiother. 2009;55(2):97-104. doi: 10.1016/s0004-9514(09)70039-x. PMID 19463080
- [Background] Jones MA, Stratton G, Reilly T, Unnithan VB. Recurrent non-specific low-back pain in adolescents: the role of exercise. Ergonomics. 2007 Oct;50(10):1680-8. doi: 10.1080/00140130701587327. PMID 17917907
- [Background] Whistance RS, Adams LP, van Geems BA, Bridger RS. Postural adaptations to workbench modifications in standing workers. Ergonomics. 1995 Dec;38(12):2485-503. doi: 10.1080/00140139508925282. PMID 8586077
- [Background] Barr KP, Griggs M, Cadby T. Lumbar stabilization: a review of core concepts and current literature, part 2. Am J Phys Med Rehabil. 2007 Jan;86(1):72-80. doi: 10.1097/01.phm.0000250566.44629.a0. PMID 17304690
- [Background] Scannell JP, McGill SM. Lumbar posture--should it, and can it, be modified? A study of passive tissue stiffness and lumbar position during activities of daily living. Phys Ther. 2003 Oct;83(10):907-17. PMID 14519062
- [Background] Mikkelsson LO, Nupponen H, Kaprio J, Kautiainen H, Mikkelsson M, Kujala UM. Adolescent flexibility, endurance strength, and physical activity as predictors of adult tension neck, low back pain, and knee injury: a 25 year follow up study. Br J Sports Med. 2006 Feb;40(2):107-13. doi: 10.1136/bjsm.2004.017350. PMID 16431995